CLINICAL TRIAL: NCT06197529
Title: Is Nociceptive Processing Evoked by Heat Homeostatically Regulated: A Contact-heat Evoked Potentials Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Daniela Montemayor Zolezzi, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CHEPS-DMZ-CNAP
Record Dates: First submitted 2023-11-22; First posted 2024-01-09 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Homeostatic Plasticity; Capsaicin; Transcranial Direct Current Stimulation
MeSH Terms: interventions — Single Person; Capsaicin; Transdermal Patch; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- S1 Homeostatic Plasticity-Pain (Experimental): Anodal tDCS CP3 1mA FP2 -1mA
  4x4 patch on the dorsum of the hand
  Interventions: Other: Homeostatic Plasticity; Drug: Topical alone (Capsaicin 8% Patch)
- S1 Homeostatic Plasticity-NoPain (Placebo Comparator): Anodal tDCS C3 1mA FP2 -1mA
  4x4 patch on the dorsum of the hand
  Interventions: Other: Homeostatic Plasticity; Other: Placebo Patch
- S1 Homeostatic Plasticity-Sham (Sham Comparator): Sham tDCS C3 FP2
  4x4 patch on the dorsum of the hand
  Interventions: Other: Placebo Patch; Other: Homeostatic Plasticity (Sham)
- M1 Homeostatic Plasticity (Active Comparator): Anodal tDCS C3 1mA FP2 -1mA
  4x4 patch on the dorsum of the hand
  Interventions: Other: Homeostatic Plasticity; Other: Placebo Patch

INTERVENTIONS:
Other: Homeostatic Plasticity — Anodal tDCS S1/M1
  Arms: M1 Homeostatic Plasticity; S1 Homeostatic Plasticity-NoPain; S1 Homeostatic Plasticity-Pain
Drug: Topical alone (Capsaicin 8% Patch) — 4x4 patch
  Other Names: Qutenza Capsaicin (8%)
  Arms: S1 Homeostatic Plasticity-Pain
Other: Placebo Patch — 4x4 patch
  Arms: M1 Homeostatic Plasticity; S1 Homeostatic Plasticity-NoPain; S1 Homeostatic Plasticity-Sham
Other: Homeostatic Plasticity (Sham) — sham Homeostatic Plasticity protocol over S1
  Arms: S1 Homeostatic Plasticity-Sham

SUMMARY:
Homeostatic plasticity is a mechanism that stabilizes neuronal activity to prevent excessive nervous system excitability. This mechanism can be investigated in humans by applying two blocks of non-invasive brain stimulation, such as transcranial direct current stimulation (tDCS).

In healthy subjects, homeostatic plasticity induction over the primary motor cortex increases the amplitude of motor-evoked potentials after the first block of excitatory tDCS, which then decreases after the second block of excitatory tDCS. However, this mechanism is impaired in chronic and experimental pain, demonstrated by an increase in excitability instead of a reversal.

The role of homeostatic plasticity mechanisms in pain is yet to be unraveled, but homeostatic plasticity may hold an important role in pain development or persistence.

Thus, the aim of this study is to investigate if the cortical nociceptive response reflected by contact heat stimulation (CHEPs) is regulated by homeostatic mechanisms. For this, homeostatic plasticity will be induced in both the primary motor (M1) and sensory cortices (S1). The first research question will explore if the contact heat evoked potentials are homeostatically regulated and if this regulation is occurring locally or globally in the cortex. Additionally, it will be investigated if and how capsaicin-induced nociception interacts and effects the homeostatic response as reflected by CHEPs.

DETAILED DESCRIPTION:
Randomized, cross-over study of four sessions

ELIGIBILITY:
Inclusion Criteria:

* Healthy right-handed men and women aged 18-60 years
* Speak, read, and understand English or Danish

Exclusion Criteria:

* Pregnant, breastfeeding, or women in childbearing age not using contraceptive methods
* Regular use of cannabis, opioids or other drugs (except contraceptives)
* Current or previous neurologic, musculoskeletal, mental, or other illnesses (e.g. brain or spinal cord injuries, degenerative neurological disorders, epilepsy, major depression, cardiovascular disease, chronic lung disease, etc.)
* Current or previous chronic or recurrent pain condition (other than low back pain in patients recruited for sub-project 6, and this item does not apply to sub-project 8)
* Current regular use of analgesic medication or other medication which may affect the trial (including paracetamol and NSAIDs) For subproject 8, chronic low back pain patients may take analgesic medication provided the dosage is stable
* Open wounds, eczema, scars, or tattoos in the area of the heat stimulation (sub-project 1)
* Lack of ability to cooperate
* Recent history of acute pain particularly in the lower limbs (unless related to low back pain in patients included in sub-project 6 or 8)
* Abnormally disrupted sleep in 24 hours preceding experiment
* Any medical or other condition (i.e. musculoskeletal, cardiorespiratory, neurological, etc.)
* Contraindications to TMS application (history of epilepsy, metal implants in head or jaw, etc.)
* Unable to answer to the "Transcranial Magnetic Stimulation Adult Safety Screen" or tDCS screening questionnaire (see Bilag_v1_06092021)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Contact Heat Evoked Potentials | Pre-patch application
  Baseline (Evoked Potentials after stimulus onset from electroencephalographic channels)
Contact Heat Evoked Potentials | 30 minutes after patch application
  Post-Patch (Evoked Potentials after stimulus onset from electroencephalographic channels)
Contact Heat Evoked Potentials | During the homeostatic plasticity protocol - 0 minutes after the first block of anodal tDCS
  Post-Priming (Evoked Potentials after stimulus onset from electroencephalographic channels)
Contact Heat Evoked Potentials | 0 minutes after homeostatic plasticity induction
  Post-HP (Evoked Potentials after stimulus onset from electroencephalographic channels)
Contact Heat Evoked Potentials | 10 minutes after the homeostatic plasticity protocol
  Post-HP+10 minutes (Evoked Potentials after stimulus onset from electroencephalographic channels)

SECONDARY OUTCOMES:
Pain Intensity After Stimulation Blocks (0-10) | 0 minutes after the first block of CHEP stimulation
  Pain intensity measured using an 11-point numeric rating scale where 0= no pain and 10 = worst imaginable pain
Pain Intensity After Stimulation Blocks (0-10) | 0 minutes after the second block of CHEP stimulation
  Pain intensity measured using an 11-point numeric rating scale where 0= no pain and 10 = worst imaginable pain
Pain Intensity After Stimulation Blocks | 0 minutes after the third block of CHEP stimulation
  Pain intensity measured using an 11-point numeric rating scale where 0= no pain and 10 = worst imaginable pain
Pain Intensity After Stimulation Blocks | 0 minutes after the fourth block of CHEP stimulation
  Pain intensity measured using an 11-point numeric rating scale where 0= no pain and 10 = worst imaginable pain
Pain Intensity After Stimulation Blocks | 0 minutes after the fifth block of CHEP stimulation
  Pain intensity measured using an 11-point numeric rating scale where 0= no pain and 10 = worst imaginable pain
Presence of Allodynia After Stimulation Blocks | 0 minutes after the first block of CHEP stimulation
  Measured with a calibrated brush for the study of dynamic mechanical allodynia (Brush-05®, Somedic SenseLab AB, Sösdala, Sweden)
Presence of Allodynia After Stimulation Blocks | 0 minutes after the second block of CHEP stimulation
  Measured with a calibrated brush for the study of dynamic mechanical allodynia (Brush-05®, Somedic SenseLab AB, Sösdala, Sweden)
Presence of Allodynia After Stimulation Blocks | 0 minutes after the third block of CHEP stimulation
  Measured with a calibrated brush for the study of dynamic mechanical allodynia (Brush-05®, Somedic SenseLab AB, Sösdala, Sweden)
Presence of Allodynia After Stimulation Blocks | 0 minutes after the fourth block of CHEP stimulation
  Measured with a calibrated brush for the study of dynamic mechanical allodynia (Brush-05®, Somedic SenseLab AB, Sösdala, Sweden)
Presence of Allodynia After Stimulation Blocks | 0 minutes after the fifth block of CHEP stimulation
  Measured with a calibrated brush for the study of dynamic mechanical allodynia (Brush-05®, Somedic SenseLab AB, Sösdala, Sweden)
Pittsburg Sleeping Quality Index | Pre-intervention and pre-patch application
  The global PSQI score ranges from 0 to 21, calculated by adding seven component scores. A global score above 5 (PSQI > 5) indicates relevant sleep disturbances or poor sleep quality (Buysse et al., 1989).
BECKS Depression Inventory | Pre-intervention and pre-patch application
  The questionnaire includes 21 items which are rated on a 4-point scale (0 to 3). The total score is calculated by adding all items. Total score values from 0-13 indicate "normal ups and downs", and scores between 14-19, 20-28, and 29-63, are interpreted as mild, moderate, and severe symptoms (Beck et al., 1996; Goldstein et al., 2013; Wang and Gorenstein, 2013).
Positive and Negative Affective Schedule - Short Form | Pre-intervention and pre-patch application
  Scores can range from 10 - 50, with higher scores representing higher levels of positive/negative affect.
State-Trait Anxiety Inventory | Pre-intervention and pre-patch application
  A 40-item questionnaire that assesses state and trait anxiety with 20 items each (Skapinakis, 2014; Spielberger et al., 1983). Each subscale (S-Anxiety and T-Anxiety) uses a 4-point Linkert scale ranging from 1 ("not at all" for S- or "almost never" for T-Anxiety) to 4 ("very much so" for S- and "almost always" for T-Anxiety). A higher scole indicates more severe anxiety with a range from 20-80.
Pain Catastrophizing Scale | Pre-intervention and pre-patch application
  This questionnaire assesses 13 items describing different thoughts and feelings which may be associated with pain. They are rated on a 5-point scale (0-5) indicating the degree to which these thoughts and feelings are present when having pain. The total score is 0-52, with a higher score indicating a higher pain catastrophizing. (Sullivan M J L, Bishop S, Pivik J. 1995)
Pain intensity (Induced by Capsaicin) | Throughout the experimental session, every 5 minutes and up to 55 minutes after patch application
  Pain intensity measured using an 11-point numeric rating scale where 0= no pain and 10 = worst imaginable pain

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Graven-Nielsen, PhD, DMSc, Study Director — Aalborg University
Locations (1):
- Aalborg University / Center for Neuroplasticity and Pain, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be available online, but the data collected can be shared upon reasonable request.

REFERENCES:
- [Background] Wittkopf PG, Larsen DB, Gregoret L, Graven-Nielsen T. Prolonged corticomotor homeostatic plasticity - Effects of different protocols and their reliability. Brain Stimul. 2021 Mar-Apr;14(2):327-329. doi: 10.1016/j.brs.2021.01.017. Epub 2021 Jan 24. No abstract available. PMID 33503491
- [Background] Wittkopf PG, Larsen DB, Graven-Nielsen T. Protocols for inducing homeostatic plasticity reflected in the corticospinal excitability in healthy human participants: A systematic review and meta-analysis. Eur J Neurosci. 2021 Aug;54(4):5444-5461. doi: 10.1111/ejn.15389. Epub 2021 Jul 30. PMID 34251703
- [Background] Wittkopf PG, Boye Larsen D, Gregoret L, Graven-Nielsen T. Disrupted Cortical Homeostatic Plasticity Due to Prolonged Capsaicin-induced Pain. Neuroscience. 2023 Nov 21;533:1-9. doi: 10.1016/j.neuroscience.2023.09.011. Epub 2023 Sep 27. PMID 37774909
- [Background] Thapa T, Graven-Nielsen T, Schabrun SM. Aberrant plasticity in musculoskeletal pain: a failure of homeostatic control? Exp Brain Res. 2021 Apr;239(4):1317-1326. doi: 10.1007/s00221-021-06062-3. Epub 2021 Feb 26. PMID 33635391
- [Background] Thapa T, Graven-Nielsen T, Chipchase LS, Schabrun SM. Disruption of cortical synaptic homeostasis in individuals with chronic low back pain. Clin Neurophysiol. 2018 May;129(5):1090-1096. doi: 10.1016/j.clinph.2018.01.060. Epub 2018 Feb 9. PMID 29472134
- [Background] Lejeune N, Petrossova E, Frahm KS, Mouraux A. High-speed heating of the skin using a contact thermode elicits brain responses comparable to CO2 laser-evoked potentials. Clin Neurophysiol. 2023 Feb;146:1-9. doi: 10.1016/j.clinph.2022.11.008. Epub 2022 Nov 24. PMID 36473333
- [Background] Lenoir C, Algoet M, Mouraux A. Deep continuous theta burst stimulation of the operculo-insular cortex selectively affects Adelta-fibre heat pain. J Physiol. 2018 Oct;596(19):4767-4787. doi: 10.1113/JP276359. Epub 2018 Sep 4. PMID 30085357